CLINICAL TRIAL: NCT06738537
Title: Patient-Centered Approach for Treatment Decisions in Mitral Valve Prolapse (PRIMARY SDM)
Brief Title: Patient-Centered Approach for Treatment Decisions in Mitral Valve Prolapse
Acronym: PRIMARY SDM
Status: Recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: West Virginia University (Other); Cedars-Sinai Medical Center (Other); The Cleveland Clinic (Other); University of Kansas Medical Center (Other); Saint Luke's Mid America Heart Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: 23-0905
Record Dates: First submitted 2024-11-08; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Mitral Valve Prolapse
Keywords: transcatheter edge-to-edge repair; surgical mitral valve repair
MeSH Terms: conditions — Mitral Valve Prolapse | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with MR: We will recruit patients with degenerative mitral regurgitation (MR) who are presenting to a surgeon or cardiologist for consultation regarding management of their valve disease.
  Interventions: Other: Focus Groups/Quantitative Survey for Patients
- Health Care Providers: We will recruit Health Care providers (cardiac surgeons and cardiologists) who evaluate and treat patients with mitral regurgitation.
  Interventions: Other: Focus Group/Quantitative Survey for HCPs
- Multidisciplinary Mitral Valve Heart Team: We will recruit members of multidisciplinary mitral valve heart teams including cardiac surgeons, cardiologists, nurses, and ancillary staff. These providers will be involved in caring for patients who presents to multidisciplinary heart teams for evaluation of their mitral valve disease.
  Interventions: Other: Qualitative Focus Group

INTERVENTIONS:
Other: Focus Groups/Quantitative Survey for Patients — 5 quantitative focus groups will be conducted with 5-10 patients each to elicit the range of outcomes patients consider important when selecting treatment options. 100 quantitative surveys to characterize how patients with severe MR prioritize outcomes when making treatment decisions.
  Groups: Patients with MR
Other: Focus Group/Quantitative Survey for HCPs — 5 quantitative focus groups will be conducted with 5-10 providers to elicit the range of outcomes providers consider important when recommending treatment options to patients. 100 quantitative surveys to characterize how providers prioritize outcomes for patients with severe MR when making treatment recommendations.
  Groups: Health Care Providers
Other: Qualitative Focus Group — Qualitative focus groups will be conducted to determine barriers and facilitators to implementing shared decision making in multidisciplinary mitral valve heart team clinics.
  Groups: Multidisciplinary Mitral Valve Heart Team

SUMMARY:
This is a qualitative and quantitative study that seeks to obtain information from patients with degenerative mitral valve prolapse and providers regarding factors important in deciding between surgical mitral valve repair (MVR) and transcatheter edge-to-edge repair (TEER). Findings from this study will provide data that can be used to develop decision aids that can assist patients in decision making between these two therapies and assist providers in integrating shared decision making the within the multidisciplinary heart valve team.

DETAILED DESCRIPTION:
Prior qualitative research in decision-making related to heart valve disease has occurred largely in transcatheter aortic valve replacement (TAVR). Among patients undergoing TAVR, physicians estimate patients' symptoms and functional status poorly both before and after treatment. Prior studies have shown that significant variability exists in outcomes most important to patients versus those most important to providers. Specifically, providers may place greater emphasis on clinical endpoints such as mortality or echocardiographic improvement in valve function whereas patients often place greater emphasis on quality-of-life outcomes such as having greater independence, feeling better, and being able to return to daily activities.

These disparities between patient and provider preference in outcomes in TAVR highlight the importance of prospectively measuring patient and provider preferences in outcomes of transcatheter edge-to-edge repair (TEER) and surgical mitral valve repair (MVR), which share similar tradeoffs in decision-making. The ongoing Percutaneous or Surgical Repair In Mitral Prolapse And Regurgitation for ≥60 Year-olds (PRIMARY) trial will compare TEER to MVR in patients with primary, degenerative MR. To allow for the creation of a decision aid that can be utilize simultaneously with completion of the parent clinical trial, the investigators seek to conduct a quantitative and quality study of patient and physician factors that influence decision-making in TEER versus MVR for degenerative mitral regurgitation.

This study will consist of prospectively conducted qualitative focus groups among patients and providers (surgeons and cardiologists) to elicit the range of outcomes when considering TEER or MVR. These data will be analyzed to develop a consolidated framework of outcomes patients and providers value. Using these data, the investigators will then create and administer a quantitative survey to characterize how patients with severe MR and their providers prioritize outcomes when making treatment decisions and recommendations. The survey will include an allocation task whereby participants will be presented with a set of alternative treatment outcomes from the qualitative surveys and components of the PRIMARY composite endpoint and asked to allocate a total of 100 points across these outcomes based on their preferences. Lastly, the investigators will identify barriers and facilitators for implementing shared decision making (SDM) in multidisciplinary mitral valve hear teams by conducting qualitative focus groups across health care provider stakeholders (e.g. surgeons, cardiologists, nurses in office). These data will be used to map workflows and identify the optimal timing and process of integrating SDM in clinical care. In addition to generating process maps, an understanding of the implementation barriers and facilitators will aid in developing an approach to create and test an implementation strategy for SDM in severe degenerative MR. Collectively, these aims lay the foundation for developing and implementing a patient centered decision aid to support SDM in the future, but also model a novel approach for implementing the results of PRIMARY into routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years and older
* Diagnosis of degenerative mitral valve regurgitation

Exclusion Criteria:

* Non-English speaking
* Unable to consent on own behalf
* Previous mitral surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe degenerative MR
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-28 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Identify outcomes most important to patients with severe degenerative MR considering TEER or MVR | 1 year
  The investigators will conduct qualitative focus groups among patients with severe degenerative MR to elicit the range of outcomes patients consider important when selecting treatment options. These data will be analyzed to develop a consolidated framework of outcomes patients value. Using these data, the investigators will then create and administer a quantitative survey to characterize how patients with severe MR prioritize outcomes when making treatment decisions.
Identify outcomes most important to healthcare providers (HCPs) in recommendingTEER or MVR | 1 year
  The investigators will conduct qualitative focus groups among cardiac surgeons, referring cardiologists, interventional cardiologists who perform TEER, and nurses involved in the care of patients with degenerative MR to characterize outcomes important to HCPs when evaluating MVR versus TEER. Using similar methods as above, the investigators will then use these data to create and administer a quantitative point allocation survey to characterize how HCPs prioritize outcomes when evaluating treatment options for severe degenerative MR patients.
Identify barriers and facilitators to implementing shared decision making (SDM) in multidisciplinary mitral valve Heart Teams | 1 year
  To support the future implementation of SDM, the investigators will evaluate the process of introducing SDM into local Heart Teams by conducting qualitative interviews across HCP stakeholders. Key stakeholders will include multidisciplinary groups of HCPs, ancillary staff, and administrators. These data will be used to map workflows and identify the optimal timing and process of integrating SDM in clinical care. In addition to generating process maps, an understanding of the implementation barriers and facilitators will aid in developing an approach to create and test an implementation strategy for SDM in severe degenerative MR.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Iribarne, MD, MS, FACC, Principal Investigator — Northwell Health
Locations (5):
- United States (5):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Saint Luke's Hospital, Kansas City, Missouri
  - Northwell Health, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - West Virginia University Medicine, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided